CLINICAL TRIAL: NCT04511871
Title: A Phase I Trial to Assess Safety, Tolerability and Anti-tumor Activity of Autologous T Cell Modified Chimeric Antigen Receptor (CAR) (CCT303-406) in Patients With Relapsed or Refractory HER2 Positive Solid Tumors
Brief Title: A Phase I Trial of CCT303-406 in Patients With Relapsed or Refractory HER2 Positive Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai PerHum Therapeutics Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCT303-406-mST01
Record Dates: First submitted 2020-08-10; First posted 2020-08-13 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumor; Gastric Cancer; Breast Cancer; Ovarian Cancer; Sarcoma
Keywords: HER2; CAR-T; Solid tumors
MeSH Terms: conditions — Stomach Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CCT303-406 (Experimental): To determine the safety, tolerability, dose-limiting toxicities (DLT) and maximum tolerated dose (MTD) of CCT303-406 cell therapy in patients with HER2-positive (IHC 3+ in ≥50% tumor cells) relapsed or refractory solid tumors.
  Dose cohorts:
  * Dose 1: 3x10^5 CCT303-406 CAR-positive T cells/kg body weight, intravenous infusion
  * Dose 2: 1x10^6 CCT303-406 CAR-positive T cells/kg body weight, intravenous infusion
  * Dose 3: 1x10^7 CCT303-406 CAR-positive T cells/kg body weight, intravenous infusion
  Interventions: Biological: CCT303-406

INTERVENTIONS:
Biological: CCT303-406 — Blood will be collected from subjects to isolate peripheral blood mononuclear cells for the production of CCT303-406. Subjects will receive the conditioning chemotherapy regimen of cyclophosphamide and fludarabine for lymphodepletion followed by a single dose of CCT303-406 via intravenous injection.

SUMMARY:
This clinical study is to investigate the safety and tolerability of CCT303-406 CAR modified autologous T cells (CCT303-406) in subjects with relapsed or refractory stage IV metastatic HER2-positive solid tumors.

DETAILED DESCRIPTION:
This is a single arm, open label, dose escalation clinical study to evaluate the safety and preliminary therapeutic efficacy of CCT303-406 cells in adult subjects with HER2 positive relapsed or refractory stage IV metastatic solid tumors.

Subjects that meet inclusion criteria with positive biopsy HER2 (IHC 3+ in ≥50% tumor cells) will receive CCT303-406 according to the 3+3 dose escalation design.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with willingness to be in the study and follow all study procedures, and capable of providing informed consent
2. Male or female aged 18-70 years
3. Patients with stage IV (according to the 8th edition of AJCC) advanced solid tumor malignancies that have failed standard treatment of relapsed or difficult-to-treat solid tumors confirmed by histology or cytology
4. At least one measurable lesion, i.e. the length of non-lymph node lesions examined according to CT cross-sectional scanning or magnetic resonance imaging (MRI), or the short diameter of the lymph node lesions is ≥15 mm according to RECIST 1.1
5. Tumors with HER2 IHC 3+ in≥50% of all tumor cells as determined by IHC according to the Breast Cancer HER2 Testing (2019 edition) and the Gastric Cancer HER2 Testing (2016 edition); For HER2 IHC 3+ tumors other than gastric and breast cancers, FISH is required to confirm HER2 expression; For relapsed patients after HER2-targeted therapies, biopsy and IHC are required to confirm HER2 expression per enrollment criteria.
6. ECOG Performance Status 0-1
7. Expected survival greater than 12 weeks
8. Adequate organ and hematopoietic system functions to meet the following requirements:

   * Hemoglobin (HGB) s 90 g/L, no blood transfusions within two weeks;
   * White blood cell (WBC) count≥2.5×109/L
   * Absolute Neutrophil Count (ANC) ≥1.5 x 109/L
   * Platelet (PLT) count ≥80-109/L
   * Total bilirubin (TBIL) ≤3.0ng/dL or ≤5 ULN
   * ALT and AST ≤5 ULN; for liver metastasis, ALT and AST ≤5 ULN
   * Creatinine (Cr) ≤1.5 x ULN; or creatinine removal rate (CrCl) ≥50 mL/min
9. LVEF≥50%
10. Serum troponin T <0.03 ng/mL
11. PT: INR < 1.7 or extended PT to normal value < 4s
12. Normal language, recognition and consciousness assessed by investigator during screening phase
13. Capable of receiving treatment and follow-up, including treatment in the clinical center;
14. Female subjects of childbearing age must take acceptable measures to minimize the likelihood of pregnancy during the trial. The results of serum or urine pregnancy test must be negative
15. Female subjects must not be in the lactation period.

Exclusion Criteria:

1. Females with pregnancy or in lactation period
2. Patients with active hepatitis B, or active hepatitis C
3. HIV positive
4. Other active infections of clinical significance
5. Patients receiving in situ surgery within 3 months
6. Patients with the following previous or accompanying diseases:

   • Patients diagnosed as severe autoimmune diseases that require long term (more than 2 months) treatment with systemic immunosuppressants (steroids), or diseases with immune-mediated symptoms, including ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus (SLE), and autoimmune vasculitis
7. Patients with ≥Grade 2 peripheral neuronal diseases (according to NCI-CTCAE v5.0)
8. Patients with any mental illness, including dementia, mental changes, which may cause difficulties understanding the informed consent and related questionnaires
9. Patients with serious uncontrollable diseases, which may interfere with the therapies in this study
10. Patients with other active malignancies in the past 5 years excluding those with completely cured basal or squamous skin cancers, superficial bladder cancers or primary breast cancers without need of follow-up treatment
11. Patients receiving systemic steroids or steroid inhalants
12. Patients who have received tumor immunotherapy (including monoclonal antibody or cell therapy) in the past 4 weeks
13. Patients allergic to immunotherapies or related drugs
14. Patients with metastatic lesions in meninges or central nervous system, or clear evidence of central nervous system diseases with continous significant symptoms in the last 6 months
15. Patients with NYHA class II heart failure, or hypertension incontrollable by standard care, or medical history of myocarditis, or heart attack within a year
16. Patients who have received or are going to receive organ transplantation
17. Patients with active bleeding
18. Patients with incontrollable pleural or abdominal fluid that needs clinical treatment or intervention
19. Patients having undergone major surgery within 4 weeks or have not fully recovered from prior surgery
20. Patients that have received radiotherapy within 4 weeks, excluding those who received local irradiation for the peripheral bone metastatic lesions for more than 2 weeks, and recovered from all acute toxicities of radiotherapy
21. Patients that have received anthracyclines within 8 weeks
22. Patients as determined by the investigators to be inappropriate for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2025-03-29 (Estimated)

PRIMARY OUTCOMES:
MTD: to determine the maximum tolerated dose of CCT303-406 | 28 days following infusion
  To assess the DLT (dose limiting toxicities) attributed to CCT303-406 per cohort and determine the RP2D (recommended phase 2 dose).

SECONDARY OUTCOMES:
ORR (overall response rate): Proportion of subjects with the best overall response (BOR) | Up to 52 weeks
  Best overall response (BOR) of subjects with PR (partial response) and CR (complete response) as determined by local investigator using RECIST 1.1
12 month survival rate | Up to 52 weeks
  The proportion of living subjects within 52 weeks of infusion
DCR: Disease control rate | Up to 52 weeks
  The proportion of subjects with CR (complete response), PR (partial response) or SD (stable disease lasting over 6 months) as determined by local investigator using RECIST 1.1.
DOR: Duration of reponse | Up to 52 weeks
  The duration of time from record of response to first progression of disease as determined by RECIST 1.1 or death date not relevant to disease progression
PFS: Progression free survival | Up to 52 weeks
  The time of disease progression by RECIST 1.1 or death since cell infusion
AE: Adverse Events | Up to 52 weeks
  The incidence, severity and duration of AE, TEAE and SAE as determined by NCI-CTCAE v5.0
The expansion over time of genetically modified CCT303-406 cells in the peripheral blood as determined by QPCR (copies/ug gDNA) | Up to 52 weeks
  PK: Pharmacokinetics
The persistence over time of genetically modified CCT303-406 cells in the peripheral blood as determined by Flow Cytometry (% CAR + cells) | Up to 52 weeks
  PK: Pharmacokinetics

OTHER OUTCOMES:
Exploration of target-efficacy correlation | Up to 52 weeks
  The correlation between levels of HER2 expression and ORR

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China